CLINICAL TRIAL: NCT03635294
Title: Multi-Omics and IPSCs to Improve the Diagnosis of Rare Intellectual Disabilities
Brief Title: Multi-Omics and IPSCs to Improve Diagnosis of Rare Intellectual Disabilities
Acronym: MIDRID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC17_0224
Record Dates: First submitted 2018-08-10; First posted 2018-08-17 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Rare Intellectual Disabilities
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample (Experimental): Blood sample for analyses
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — combining genomics, transcriptomics, metabolomics and morphological analyses performed on induced pluripotent stem cell (iPSC)-derived neural cells

SUMMARY:
Background Genetic factors play a major role in intellectual disability (ID) but the underlying cause is not determined in many cases.

This proposal is the continuation of the previous interregional project HUGODIMS, the aim of which was to perform whole exome sequencing (WES) in 69 thoroughly selected simplex ID parent-child trios. Thanks to HUGODIMS consortium, the underlying genetic cause of ID was determined or highly suspected in 48 cases (69.5%) and 7 novel ID genes were identified.

Hypothesis Investigators hypothesize that an approach combining genomics, transcriptomics, metabolomics and morphological analyses performed on induced pluripotent stem cell (iPSC)-derived neural cells would improve diagnosis of ID. The current proposal is therefore a proof-of concept project aiming at assessing the relevance and effectiveness of this multi-omics approach.

Aims and Methods Ten individuals with ID recruited through HUGODIMS, in whom WES have failed to identify pathogenic variants will be included.

The workflow is the following:

1. Whole genome sequencing (WGS) (Nantes) of these 10 negative trios.
2. Bio-informatics analyses
3. In 3 WGS negative cases, 3 positive controls bearing distinct mutations in CAMK2a (a novel ID gene identified thanks to HUGODIMS), and 3 healthy negative controls:

   1. Derivation of induced pluripotent stem cell (iPSC)-derived neural progenitors (iPSC core facility at Nantes)
   2. Targeted and non-targeted metabolomics analyses performed on iPSC-derived neuronal cells (Angers)
   3. RNA sequencing performed on the 9 cell lines (Rennes)
   4. Morphological analyses of differentiated neuronal cell lines derived from 3 affected individuals and 3 positive controls bearing CMK2a mutations (Tours)
   5. Integration and validation of data from multi-omics and morphological approaches

Expected results and impact Investigatrors expect that this approach combining multi-omics and iPSC will help to improve diagnosis and understanding of genetic ID of unknown cause

ELIGIBILITY:
Inclusion Criteria:

* 3 Whole Genome Sequencing negative cases
* 3 positive controls bearing distinct mutations in CAMK2a

Exclusion Criteria:

* no informed consent/refusal

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the relevance and effectiveness of a multi-omics approach to the diagnosis of ID of unknown genetic origin. | Day 1
  Whole genome sequencing : de novo variants in non-coding regions of the genome, WGS will be performed using the HiSeq X Five System 5; Bionformatics analysis of WGS data; neuronal progenitors derived from iPSC

SECONDARY OUTCOMES:
The assessment of metabolomics consequences of CAMK2a mutations in human neuronal progenitors and differentiated neuronal cell lines | Day 1
  Coupled to high-resolution mass spectrometry ; Transcriptomics analyses: quality of the RNA will be evaluated with the Bioanalyzer (Agilent) on the basis of the RIN (RNA integrity number) as well as by taking into account the DV200, i.e. the percentage of RNA fragments with more than 200 nucleotides Non-targeted metabolomic analyses will be performed using a method based on ultra-high-performance liquid chromatography Flow injection analysis-tandem mass spectrometry for quantifying acylcarnitines, glycerophospholipids, sphingolipids and sugar, whereas liquid chromatography
The assessment of morphological consequences of CAMK2a mutations in human neuronal progenitors and differentiated neuronal cell lines | Day 1
  immunocytochemistry and protein expression approaches using confocal microscopy and Western blotting with antibodies specific for proteins expressed in neurons (MAP2, Tubulin beta 3, PSD95, SNAP25), astrocytes (GFAP) or oligodendrocytes (Gal-C)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Angers, Angers
  - HCL Lyon, Bron
  - CHU de Bourgogne, Dijon
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No